CLINICAL TRIAL: NCT04161404
Title: A Phase 1, Open Label, Randomized, Three-Period, Crossover, Single Dose Oral Administration Of Andrographis Paniculata And Metformin Clinical Trial In Healthy Volunteers Under Fasting Condition
Brief Title: Pharmacometabolomics of Andrographis Paniculata And Metformin In Healthy Volunteers Under Fasting Condition
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P1-PKPD-Metabolomic
Record Dates: First submitted 2019-11-04; First posted 2019-11-13 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Pharmacokinetics; Molecular Mechanisms of Pharmacological Action
Keywords: Pharmacometabolomic; Metformin; Andrographis paniculata; Metabolomics; Phase 1; Healthy volunteers; Herbal Medicine
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Open label, block-randomized, three-period, crossover, single dose oral administration of investigational products. Subjects will undergo at least 7 days washout period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Period 1 (Experimental): Subjects will randomized to either of the intervention drug in a ratio of 1:1:1 following three period, cross-over study design.
  Interventions: Drug: Brand name: Andrographis paniculata (Shine Hempedu Bumi) 1000mg capsules; Drug: Brand name: Andrographis paniculata (Shine Hempedu Bumi) 2000mg; Drug: Metformin (Glucophage) 1000mg
- Period 2 (Experimental): Subjects will randomized to either of the intervention drug in a ratio of 1:1:1 following three period, cross-over study design.
  Interventions: Drug: Brand name: Andrographis paniculata (Shine Hempedu Bumi) 1000mg capsules; Drug: Brand name: Andrographis paniculata (Shine Hempedu Bumi) 2000mg; Drug: Metformin (Glucophage) 1000mg
- Period 3 (Experimental): Subjects will randomized to either of the intervention drug in a ratio of 1:1:1 following three period, cross-over study design.
  Interventions: Drug: Brand name: Andrographis paniculata (Shine Hempedu Bumi) 1000mg capsules; Drug: Brand name: Andrographis paniculata (Shine Hempedu Bumi) 2000mg; Drug: Metformin (Glucophage) 1000mg

INTERVENTIONS:
Drug: Brand name: Andrographis paniculata (Shine Hempedu Bumi) 1000mg capsules — Andrographis paniculata or hempedu bumi capsule is a traditional medicinal product registered under Ministry of Health Malaysia for general wealth being. It is traditionally used for anti-diabetic, anti-bacterial, anti-pyretic, anti-malarial, anti-inflammatory, antidiarrhoeal and other effects.
  Other Names: Product name: Shine Hempedu Bumi
Drug: Brand name: Andrographis paniculata (Shine Hempedu Bumi) 2000mg — Andrographis paniculata or hempedu bumi capsule is a traditional medicinal product registered under Ministry of Health Malaysia for general wealth being. It is traditionally used for anti-diabetic, anti-bacterial, anti-pyretic, anti-malarial, anti-inflammatory, antidiarrhoeal and other effects.
  Other Names: Product name: Shine Hempedu Bumi
Drug: Metformin (Glucophage) 1000mg — Metformin is an oral glucose-lowering drug of the biguanides class. Drug: Period 1 Subjects
  Other Names: Brand name: Glucophage

SUMMARY:
This study is a phase 1, open label, randomized, three-way crossover, single dose, oral- administration of Andrographis paniculata and Metformin in healthy volunteers under fasting condition. The study will demonstrate the pharmacokinetics profile and pharmacodynamic through metabolic pathway analysis for Andrographis paniculata and Metformin.

DETAILED DESCRIPTION:
This is a phase 1, open label, randomized, three period, crossover, single dose oral administration of Andrographis Paniculata 1000mg, 2000mg and Metformin 1000mg clinical trial in healthy volunteers under fasting condition. Approximately 18 healthy volunteers will be enrolled into this study.

The healthy volunteers will be screened for inclusion and exclusion criteria. Eligible subjects will be enrolled into either Metformin 1000mg tablet, Andrographis Paniculata 1000mg or 2000mg capsule in a ratio of 1:1:1 in period 1 for single dose oral administration. Subjects will then undergo a washout period of at least 7 days. After the washout period, subjects will crossover over to another investigational product according to the randomization sequence.

Subjects will fast overnight prior to dosing. The volunteers will be admitted to Clinical Investigation Center ward at 7 am in the morning and will confine in air-conditioning environment with beds and chairs. The means during the stay at CIC ward will be provided to the subjects. The dosing will be performed at 8am. A series of plasma will be collected at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12 and 24 hours post-dose. Urine samples will be collected at 0, 0-4 hours, 4-8 hours and 8-12 hours.

A safety follow-up call will be made to subjects to record any adverse events that occurred post-dosing within 1 week.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: male
2. 18 to 45 years of age (inclusive both)
3. BMI 18.5 - 29.5 kg/m2 (inclusive both) with minimum weight of 50kg
4. Non-smokers
5. Legible and willing to provide written informed consent.

Exclusion Criteria:

1. Volunteers suffering from any chronic illness such as arthritis, asthma, etc.
2. History of pre-existing bleeding disorder.
3. Clinically relevant abnormalities in the results of the laboratory screening evaluation.
4. Clinically significant abnormal electrocardiogram (ECG).
5. Positive HIV or positive hepatitis B or C in screening test or no known other hepatitis infection.
6. History of significant blood loss due to any reason, including blood donation in the past 3 months.
7. Participation in any study within past 3 months
8. History of alcohol or drug abuse
9. History of consumption of prescribed medication since last 14 days or Over-the-counter medication/ herbal remedies since last 7 days before beginning of the study.
10. Systolic blood pressure less than 100 mmHg or more than 139 mmHg and diastolic blood pressure less than 60 mmHg or more than 89 mmHg.
11. Pulse rate less than 60/minutes or more than 100/minute unless deem not clinically significant by investigator.
12. Oral temperature more than 37.5 degree Celsius.
13. History of allergy to the investigational product or any drug chemically similar to the drug under investigation.
14. Recent history of kidney or liver dysfunction.
15. Volunteers suffering from any psychiatric (acute or chronic) disorder.
16. Existence of any surgical or medical condition, which, in the judgment of the chief investigator and/or clinical investigator/physician, might interfere with the absorption, distribution, metabolism or excretion of the drug or likely to compromise the safety of volunteers.
17. Inability to communicate or co-operate.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-08-21 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of Andrographis paniculata | 0-24 hours
  Area under the plasma concentration curve of Andrographis paniculata from administration to 24 hours
Cmax of Andrographis paniculata | 0-24 hours
  Maximum plasma concentration of Andrographis paniculata after single dose oral administration.
Tmax of Andrographis paniculata | 0-24 hours
  Time until Cmax of Andrographis paniculata is reached after single dose oral administration.
Area under the plasma concentration-time curve (AUC) of Metformin | 0-24 hours
  Area under the plasma concentration curve of Metformin from administration to 24 hours
Cmax of Metformin | 0-24 hours
  Maximum plasma concentration of Metformin after single dose oral administration.
Tmax of Metformin | 0-24 hours
  Time until Cmax of Metformin is reached after single dose oral administration.

SECONDARY OUTCOMES:
Metabolic pathway of Andrographis paniculata | 24 hours
  Pre-dose and post-dose samples will be analysed using LCMSMS. Normalization, log-transformation and center scaling will then apply to batches of chromatograms. Global metabolomics analyses will be performed to identify significant endogenous metabolites between post-dose and pre-dose samples using T-Test, Principal Component Analysis, Partial Least Square Discriminant Analysis. Annotations of significant compounds will be perform using METLIN database. The significant compounds will lead to prediction of relevant metabolomic pathway from Human Metabolome Database/ Kyoto Encyclopedia of Gene and Genome pathway for Andrographis paniculata.
Metabolic pathway of Metformin | 24 hours
  Pre-dose and post-dose samples will be analysed using LCMSMS. Normalization, log-transformation and center scaling will then apply to batches of chromatograms. Global metabolomics analyses will be performed to identify significant endogenous metabolites between post-dose and pre-dose samples using T-Test, Principal Component Analysis, Partial Least Square Discriminant Analysis. Annotations of significant compounds will be perform using METLIN database. The significant compounds will lead to prediction of relevant metabolomic pathway from Human Metabolome Database/ Kyoto Encyclopedia of Gene and Genome pathway for Metformin.
Adverse drug reaction | 3 weeks
  Number of subjects with adverse drug reaction

CONTACTS AND LOCATIONS:
Overall Officials: Khim Boon Tee, Principal Investigator — University of Malaya
Locations (1):
- Clinical Investigation Centre, University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
We will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions by Medical Research Ethics Committee, University Malaya Medical Centre.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The information is available approximately in December 2020 or when the study is published. The data is available for 2 years.
Access Criteria: Kindly email to Tee Khim Boon for the above information.

REFERENCES:
- See also: Medical Research Ethics Committee, University Malaya Medical Centre — http://www.ummc.edu.my/research/research_ethics.asp?keyid=